CLINICAL TRIAL: NCT02056470
Title: A Prospective, Multicenter, Single Arm Adaptive-Design Study to Evaluate the Safety, Functionality, and the Quality of Life of Patients Who Receive the Freedom Total Knee ® System
Brief Title: Evaluate the Safety, Functionality, and the Quality of Life of Patients Who Receive the Freedom Total Knee ® System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxx Orthopedics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO-U-101A
Record Dates: First submitted 2014-02-03; First posted 2014-02-06 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Knee Joint Pain
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Freedom Total Knee Replacement (Experimental): Freedom Total Knee
  Interventions: Device: Freedom Total Knee; Device: Total Knee Replacement; Device: Freedom Total Knee System

INTERVENTIONS:
Device: Freedom Total Knee — The Freedom Total Knee System is being implanted in subjects suitable for a total knee replacement
  Other Names: Freedom Total Knee System
Device: Total Knee Replacement — total Knee replacement implant
  Other Names: Freedom Knee
Device: Freedom Total Knee System — Total Knee replacement implant
  Other Names: Freedom Knee

SUMMARY:
Assess the safety and functionality of the Freedom Knee® system through a multi-center clinical trial. Study endpoints include a comparison of Pre-Surgery versus Post-Surgery data for:

1. Range of Motion
2. Quality of Life measurements using Knee Society Scale (KSS)
3. Survivorship as defined by 'No Revision' of baseline implant
4. Quality of Life measurements using the WOMAC Score

DETAILED DESCRIPTION:
The clinical study will involve a series of evaluations performed by your surgeon. These examinations are consistent with the normal surgeon care as part of Total Knee Replacement surgery. The study objective is to assess the safety, functionality, and survivorship of the Freedom Knee System through a multi-center clinical trial. Study endpoints include a comparison of Pre-Surgery (baseline) versus Post-Surgery data for Range of Motion and Flexion, Quality of Life (KSS), and survivorship (defined by 'no revisions'). Additionally, the structural integrity will be evaluated based on the x-ray performed 36-months after knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 40-80 years of age
* Patients requiring knee prosthesis, and have been evaluated as appropriate candidates for aTKA by their orthopedic surgeon
* Patients who understand the conditions of the study and are willing and able to comply with the post-operative scheduled clinical and the prescribed rehabilitation

Exclusion Criteria:

* Previous major knee replacement of the affected knee joint
* Other significant disabling problems from the muscular-skeletal system than in the knees (i.e muscular dystrophy, polio, nueropathic joints)
* Obese patients where obesity is severe enough to affect subject's ability to perform activities of daily living (body mass index, kg/m2: BMI > 35)
* Patients who are found to be non-compliant by their physician
* Patients with or having; malignancy - active malignancy, active or suspected infection, Paget's disease, renal osteodystrophy, immunologically suppressed, sickle cell anemia, and systemic lupus erythmatosus.
* The patient has a neuromuscular or neurosensory deficit.
* Female patients planning a pregnancy during the course of the study.
* Patients, who are mentally incompetent or are unlikely to be compliant with the prescribed post-operative routine and follow-up evaluation schedule.
* Varus or valgus deformity > 20 degrees

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Assess the safety and functionality of the Freedom Knee® system through a multi-center clinical trial | 3 years
  The study is hoping to assess the safety of the implant by looking at the incident of revisions to the implant post surgery up to and including 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Eberle, Study Director — Director, Clinical Affairs
Locations (1):
- Maxx Ortho, Norristown, Pennsylvania, United States